CLINICAL TRIAL: NCT00993317
Title: A Phase III Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, 24-week Study to Assess the Efficacy and Safety of Certolizumab Pegol as Additional Medication to MTX in Patients With Active Rheumatoid Arthritis Who Have an Incomplete Response to Methotrexate
Brief Title: A Study of CDP870 as Add-on Meditation to Methotrexate (MTX) in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101-KOA-0801i
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Rheumatoid Arthritis
Keywords: CDP870; Korea; CIMZIA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo of CDP870+MTX (Placebo Comparator)
  Interventions: Drug: Placebo of CDP870; Drug: Methotrexate
- CDP870 200mg+MTX (Experimental)
  Interventions: Drug: CDP870 200mg; Drug: Methotrexate

INTERVENTIONS:
Drug: Placebo of CDP870 — Given every 2 weeks until Week22 (SC)
  Arms: Placebo of CDP870+MTX
Drug: CDP870 200mg — 400mg CDP870 given at Week0, 2, 4 and thereafter 200mg CDP870 given every 2 weeks until Week 22(SC)
  Other Names: CIMZIA
  Arms: CDP870 200mg+MTX
Drug: Methotrexate — Received treatment with Methotrexate(MTX)for at least 24 weeks prior to the Baseline Visit.
  The dose and route of administration of MTX had to have been stable for at least 8 weeks prior to the Baseline Visit. The minimum stable dose of MTX allowed is 10mg weekly.

SUMMARY:
The objective of this trial is to compare the efficacy of Certolizumab (CZP) (CDP870) in combination with Methotrexate (MTX) to MTX alone in the treatment of signs and symptoms in patients with active rheumatoid arthritis (RA) who are incomplete responders to MTX.

ELIGIBILITY:
Inclusion Criteria:

* Adult-onset RA of at least 6 months but not longer than 15 years in duration as defined by the 1987 American College of Rheumatology classification criteria
* Active RA disease as defined by at least 9 tender joints and 9 swollen joints, ESR of 30 mm/hour or CRP of 1.5 mg/dL
* MTX (with or without folic acid) for at least 24 weeks prior to the Baseline visit, The dose of MTX and route of administration must have been stable for at least 8 weeks prior to the baseline visit. The minimum stable dose of MTX allowed is 10 mg weekly.

Exclusion Criteria:

* Any other inflammatory arthritis (e.g., psoriatic arthritis, ankylosing spondylitis or reactive arthritis)
* Secondary, non-inflammatory type of arthritis (eg, osteoarthritis, fibromyalgia)
* NYHA (New York Heart Association) Class III or IV congestive heart failure
* current or history of, tuberculosis
* history of chronic infection, recent serious or life-threatening infection (within 24 weeks , including herpes zoster), or any current sign or symptom that may indicate an infection (e.g., fever, cough)
* High risk of infection
* Have received any experimental non-biological therapy, within or outside a clinical trial in the 12 weeks prior to Baseline
* Have received previous B-cell therapy (eg. Rituximab)
* Have received any other biological therapy for RA within 24 weeks prior to Baseline visit, except for etanercept where a three month washout prior to baseline visit is acceptable
* Have received previous treatment with a biological therapy for RA that resulted in a severe hypersensitivity reaction or an anaphylactic reaction
* Failed to respond to previous treatment with an anti-TNF drug
* Female breast feeding, pregnant or plan to become pregnant during the trial or for 12 weeks following the last dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-kon Lee, MD. PhD, Principal Investigator — Severance Hospital
Locations (15):
- South Korea (15):
  - Kyungpook National University Hospital, Daegu
  - Catholic University Hospital of Daegu, Daegu
  - Eulji University Hospital, Daejeon
  - Inha University Hospital, Inchon
  - Chonnam National University Hospital, Kwangju
  - Pusan National University Hospital, Pusan
  - Yonsei University Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Catholic University of Korea ST.Mary's Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hanyang Universoty Hospital, Seoul
  - KonKuk University Medical Center, Seoul
  - Seoul national univeristy, Seoul
  - Ajou University Hospital, Suwon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period : from 03 Nov 2009 to 16 Dec 2010 Types of location : clinic of rheumatology
Groups:
- Placebo of CDP870+MTX: 0.9% saline solution (preservative free) given as two 1ml injections of PFS at Baseline, Weeks 2 and 4, then every two weeks given as one 1ml injection of PFS.
- CDP870 200mg+MTX: Certolizumab pegol for subcutaneous injection is supplied in a 1 ml pre-filled syringe (PFS) for single use at dosage strength of 200 mg/ml.
Period: Overall Study
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Started | 42 | 85
Completed | 21 | 60
Not Completed | 21 | 25
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 18 | 18
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Investigator's opinion | 0 | 1
Not completed — Early study termination at the site | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX | Total
Number analyzed (Participants) | 42 | 85 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 72 | 110
  >=65 years | 4 | 13 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 75 | 112
  Male | 5 | 10 | 15
Disease Duration [Mean (Standard Deviation); unit: years] | 6.0 (5.1) | 6.4 (4.2) | 6.3 (4.5)
Concomitant MTX dose [Mean (Standard Deviation); unit: mg/week] | 13.6 (2.8) | 13.4 (2.5) | 13.5 (2.6)
Number of previous disease-modifying anti-rheumatoid drugs (DMARDs) [Mean (Standard Deviation); unit: drugs/participants] | 3.2 (1.5) | 3.3 (1.3) | 3.3 (1.4)
Tender/Painful Joint Count [Mean (Standard Deviation); unit: Joints/participants] — Tender/Painful joint count range from 0-68
  Joints/participants | 25.05 (14.61) | 25.04 (14.44) | 25.04 (14.44)
Swollen Joint Count [Mean (Standard Deviation); unit: Joints/participants] — Swollen joint count range from 0-66
  Joints/participants | 17.31 (11.18) | 15.96 (8.86) | 16.41 (9.66)
Health Assessment Questionnaire Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: scores on a scale] — Total Scale Range: 0(Minimum)-3(Maximum) Lower values represent a better outcome.
  scores on a scale | 1.53 (0.74) | 1.43 (0.67) | 1.46 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: ACR20 Responses at Week 24
Description: Achieving ACR20 means 20% or greater improvement in the number of tender joints, a 20% or more improvement in the number of swollen joints and a 20% or greater improvement in at least three of the five remaining core set measures: Patient's and physician's global assessments, Patient's assessment of pain, disability index based on the Health Assessment Questionnaire and C-reactive Protein.
Time Frame: Week 24
Population: Full Analysis Set (FAS) Population The full set population will consist of all the subjects who were randomized and treated with the drug and received the primary efficacy evaluation at baseline. In the case of dosing administration error, analyses on the FAS population will be conducted according to the drug the subjects were randomized to.
Measure: Number; unit: participants
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Number analyzed (Participants) | 40 | 81
participants | 11 | 54 [2.291 to 12.137]

2. Secondary Outcome: ACR 20 Responses at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: FAS population
Measure: Number; unit: participants
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Number analyzed (Participants) | 40 | 81
participants | 15 | 52

3. Secondary Outcome: ACR50 Responses at Week 12
Description: Achieving ACR50 means 50% or greater improvement in the number of tender joints, a 50% or more improvement in the number of swollen joints and a 50% or greater improvement in at least three of the five remaining core set measures: Patient's and physician's global assessments, Patient's assessment of pain, disability index based on the Health Assessment Questionnaire and C-reactive Protein.
Time Frame: Week 12
Population: FAS population
Measure: Number; unit: participants
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Number analyzed (Participants) | 40 | 81
participants | 5 | 21

4. Secondary Outcome: ACR70 Responses at Week 12
Description: Achieving ACR70 means 70% or greater improvement in the number of tender joints, a 70% or more improvement in the number of swollen joints and a 70% or greater improvement in at least three of the five remaining core set measures: Patient's and physician's global assessments, Patient's assessment of pain, disability index based on the Health Assessment Questionnaire and C-reactive Protein.
Time Frame: Week12
Population: FAS population
Measure: Number; unit: participants
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Number analyzed (Participants) | 40 | 81
participants | 0 | 11

5. Secondary Outcome: ACR50 Responses at Week 24
Time Frame: Week 24
Population: FAS population
Measure: Number; unit: participants
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Number analyzed (Participants) | 40 | 81
participants | 8 | 35

6. Secondary Outcome: ACR70 Responses at Week24
Time Frame: Week 24
Population: FAS population
Measure: Number; unit: participants
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Number analyzed (Participants) | 40 | 81
participants | 1 | 14

7. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: Range of HAQ-DI score: 0-3 This outcome measures changes of HAQ-DI score at Week 24 from Baseline. Lower score of HAQ-DI represents a better outcome.
Time Frame: Baseline and Week 24
Population: FAS population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Number analyzed (Participants) | 40 | 81
scores on a scale | -0.17 (0.70) | -0.54 (0.51)

ADVERSE EVENTS:
Time Frame: 36weeks
Arm/Group | Placebo of CDP870+MTX | CDP870 200mg+MTX
Serious Adverse Events (participants affected / at risk) | 0/42 | 8/85
Other Adverse Events (participants affected / at risk) | 21/42 | 52/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo of CDP870+MTX (N=42) | CDP870 200mg+MTX (N=85)
Tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular spasm (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo of CDP870+MTX (N=42) | CDP870 200mg+MTX (N=85)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 12 (12)
Nasopharyngitis (Infections and infestations) | 4 (4) | 10 (14)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No